CLINICAL TRIAL: NCT03542045
Title: A Prospective Single-arm Multicenter Study to Evaluate Clinical Performance of Cemented ATTUNE® Knee System in Primary Total Knee Arthroplasty
Brief Title: China ATTUNE® Study
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: DPS-201701
Record Dates: First submitted 2018-04-10; First posted 2018-05-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Cemented ATTUNE® Knee System — This product is for total knee arthroplasty. Four implant configurations are permitted: Cruciate Retaining Fixed Bearing (CR FB), Cruciate Retaining Rotating Platform (CR RP), Posterior Stabilizing Fixed Bearing (PS FB) and Posterior Stabilizing Rotating Platform (PS RP)

SUMMARY:
The study was designed as prospective, single-arm, multi-center which was intended to broadly capture all patients as the technology is adopted.

DETAILED DESCRIPTION:
The primary objective is to evaluate the implant survivorship of ATTUNE primary, cemented Knee system in Chinese patients using Kaplan Meier Survivorship at 2 yrs. The subject population is male and female subjects who are candidates for primary, total knee arthroplasty between 18 and 80 years of age, inclusive, willing to consent with indications consistent with the Instructions for Use. A total of 120 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Subjects with Osteoarthritis (OA), post-trauma arthritis.
2. Subject is male or female and between the ages of 18 and 80 years old, inclusive.
3. Subject requires a primary total knee replacement with or without un-resurfaced patella and is considered by the Investigator to be suitable for the specific knee prosthesis identified in the protocol.
4. Subject requires unilateral knee replacement or the first knee with ATTUNE system during the study will be enrolled for bilateral knee replacement.
5. Subject, or with the aid of a family member, is able to understand the Informed Consent Document and patient questionnaires.
6. Subject, with the aid of a family member as needed, has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to the Sponsor.
7. Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.

Exclusion Criteria:

1. The Subject has, in the opinion of the Investigator, an existing condition that would compromise their participation and follow-up in this study, e.g. living in distant areas or having difficulty to return to the site, incooperative to surgeons' medical instructions and suggestions.
2. The Subject is a woman who is pregnant or lactating.
3. The Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect follow-up care or treatment outcomes.
4. The Subject has participated in a clinical investigation with an investigational product in the last 3 months that could impact/affect the outcome of the current procedure and follow-ups judged by the investigator.
5. The Subject has previous prosthetic knee replacement (any type including unicompartmental, total knee arthroplasty, patellofemoral arthroplasty or ipsilateral Upper Tibial Osteotomy (UTO)/ High Tibial Osteotomy (HTO)) of the affected knee or a previous patellectomy.
6. Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot disease, avascular necrosis).
7. The Subject requires a device not specified in the protocol or the surgeon determines that the ATTUNE Knee System is not a suitable treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female Subjects who are candidates for primary, total knee arthroplasty between 18 and 80 years of age, inclusive, willing to consent with indications consistent with the Instructions for Use.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Implant survivorship. | postoperatively 2 years.
  To evaluate the implant survivorship of ATTUNE primary, cemented Knee system in Chinese patients using Kaplan Meier Survivorship at 2 yrs.

SECONDARY OUTCOMES:
Knee society score (KSS) 2011-surgeon portion at post-operative 2 years compared to pre-op baseline. | pre-operative and post-operative 2 years.
  Questionnaire.
Knee injury and Osteoarthritis Outcome Score (KOOS) at postoperative 2 years compared to pre-op baseline. | Pre-operative baseline and post-operative 2 years.
  Questionnaire.
Euro Quality of life five Dimensions questionnaire five level (EQ5D-5L) at postoperative 2 years compared to pre-op baseline. | Pre-operative and post-operative 2 years.
  Questionnaire.
Knee society score (KSS) 2011-patient portion at post-operative 2 years compared to pre-op baseline. | Pre-operative baseline and post-operative 2 years.
  Questionnaire.
Adverse events and serious adverse events. | Up to post-operative 2 years.
  Type and frequency of adverse events and serious adverse events.
Implant survivorship. | Post-operative 1 year.
  Kaplan Meier Survivorship at 1 year.
Health economy. | Post-operative 2 years.
  Patient total charges in hospital.
Length of hospital stay. | Through hospitalization for primary surgery, an average of 2 weeks.
  Hospitalization duration for primary surgery.
Destination status. | At discharge of primary surgery, an average of post-operative 7 days.
  Home or rehabilitation department/secondary care facility/nursing facility.

OTHER OUTCOMES:
Knee Society Score (KSS) 2011-surgeon portion at post-operative 6 weeks, 6 months and 1 year compared to pre-op baseline. | Pre-operative baseline, post-operative 6 weeks, 6 months, and 1 year.
  Questionnaire.
Knee injury and Osteoarthritis Outcome Score (KOOS) at postoperative 6 weeks, 6 months, 1 year compared to pre-op baseline. | Pre-operative baseline, post-operative 6 weeks, 6 months and 1 year.
  Questionnaire.
Euro Quality of life five Dimensions questionnaire five level (EQ5D-5L) at postoperative 6 weeks, 6 months, 1 year compared to pre-op baseline. | Pre-operative baseline, post-operative 6 weeks, 6 months and 1 year.
  Questionnaire.
Knee society score (KSS) 2011-patient portion at post-operative 6 weeks, 6 months, 1 year compared to pre-op baseline. | Pre-operative baseline, post-operative 6 weeks, 6 months and 1 year.
  Questionnaire.
Radiographic evaluation. | Immediate post operation, post-operative 6 weeks and 1 year.
  Radiographic evaluation at immediate post operation and 6 weeks, 1 year visit.

CONTACTS AND LOCATIONS:
Overall Officials: Shudong Zhang, Principal Investigator — Yantaishan Hospital
Locations (1):
- Yantaishan Hospital, Yantai, Shangdong, China